CLINICAL TRIAL: NCT05734586
Title: Feasibility Study of Screening for Sarcopenic Dysphagia and the Implementation of Measures to Prevent Its Complications in Geriatric or Institutionalized Patients Aged ≥ 70 Years.
Brief Title: Screening for Sarcopenic Dysphagia and the Implementation of Measures to Prevent Its Complications in Geriatric Patients [DYSPHAGING-PILOT]
Acronym: DYSPHAGING-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0474
Record Dates: First submitted 2023-01-27; First posted 2023-02-21 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Swallowing Disorder; Sarcopanic Dysphagia
Keywords: Prevention; Nutrition; Re-education
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DYSPHAGING Interventional group (Other): * Step 1: delivery of the EAT-10 questionnaire for swallowing disorders screening;
  * Step 2: in case of EAT≥2 score, immediate implementation of upper airway protection measures in 3 areas:
    1: Postural adjustments; 2 : Hygienic and dietary rules ; 3: Food textures The hypothesis is that allied health professionals in acute geriatric wards, rehabilitation units, and Long Term Care Units are able to implement the current recommendations for screening for sarcopenic dysphagia and to implement preventive measures but in a systematic way.
  Patient characteristics will be collected at each site at the end of the study by a clinical research assistant based on their medical records.
  At the end of the study, each allied health professionals who has been involved in the care of at least one patient will fill out a satisfaction questionnaire.
  Interventions: Other: EAT-10 (Eating assessment Tool) screening questionnaire; Procedure: Protective measures for the upper airways

INTERVENTIONS:
Other: EAT-10 (Eating assessment Tool) screening questionnaire — After inclusion, issuance of the EAT-10 screening questionnaire for swallowing disorders by the healthcare team
Procedure: Protective measures for the upper airways — In the event of an EAT ≥2 score, immediate implementation or within three days by the healthcare team of protective measures for the upper airways in 3 sectors:
  1: Postural maneuvers; 2: Hygienodietetic rules; 3: Food textures

SUMMARY:
Sarcopenic dysphagia is described as a swallowing disorder caused by a loss of muscle mass and strength, sarcopenia. It induces chronic complications like micro-inhalations and the worsening of chronic undernutrition, according to a vicious circle. Awareness of the high prevalence of sarcopenic dysphagia and its serious consequences among elderly people with disabilities and hospitalized patients is recent, which explains the low rate of screening in the population concerned. In this context, methods of prevention, evaluation and intervention of sarcopenic dysphagia adapted to the most exposed population are needed.

Two European learned societies have developed recommendations that include increased awareness of swallowing disorders, the use of screening scores, preventive measures, diagnostic standardization, and implemented interventions (rehabilitation, textural adaptation, etc.). In order to respect these recommendations, a pedagogical sheet, entitled DYSPHAGING was elaborated within our unit in a multiprofessional way in 4 steps (1 - Screen; 2 - Protect; 3 - Confirm; 4 - Rehabilitate).

This feasibility study aims to evaluate the rate of completion and the conditions for implementing steps 1 and 2 in hospital and institutional care units.

DETAILED DESCRIPTION:
Sarcopenic dysphagia is described as a swallowing disorder caused by a loss of muscle mass and strength, sarcopenia. It induces chronic complications like micro-inhalations and the worsening of chronic undernutrition, according to a vicious circle. Awareness of the high prevalence of sarcopenic dysphagia and its serious consequences among elderly people with disabilities and hospitalized patients is recent, which explains the low rate of screening in the population concerned. In this context, methods of prevention, evaluation and intervention of sarcopenic dysphagia adapted to the most exposed population are needed.

Two European learned societies have developed recommendations that include increased awareness of swallowing disorders, the use of screening scores, preventive measures, diagnostic standardization, and implemented interventions (rehabilitation, textural adaptation, etc.). In order to respect these recommendations, a pedagogical sheet, entitled DYSPHAGING was elaborated within our unit in a multiprofessional way in 4 steps (1 - Screen; 2 - Protect; 3 - Confirm; 4 - Rehabilitate).

This feasibility study aims to evaluate the rate of completion and the conditions for implementing steps 1 and 2 in hospital and institutional care units.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 70 years,
* Patient affiliated to a social security system,
* Patient hospitalized in the health sector or in a medico-social institute,
* Patient informed of the study (information leaflet provided) and having orally signified their consent to inclusion in the study.
* Patient under legal protection, guardianship or curatorship,

Exclusion Criteria:

* Patient unable to feed orally,
* Patient with an active pathology responsible for acute swallowing disorders (< 3 months) (neurodegenerative pathology with predominant motor impairment such as Charcot's disease, stroke, ENT disease).
* Patient unable to answer the questionnaire.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of complete achievement of steps 1 and 2 | Three days
  The judgment criterion is validated if
  1. Stage 1 is performed and the EAT-10 < 2 or if
  2. Stage 1 is performed with an EAT-10 ≥ 2 and stage 2 is performed within 3 days after stage 1

SECONDARY OUTCOMES:
Percentage of eligible patients refusing to participate in the study | 18 months
  Number of eligible patients who refused to participate in the study
Age, gender, comorbidities (CIRS-G), autonomy (ADL, IADL), co-medications | 19 months
  Patient characteristics will be collected at each site at the end of the study by a clinical research assistant based on their medical records.
Rate of partial completion of the protocol | 19 months
  Proportion of non-performance of step 1 and/or step 2 within the time limit. Proportion of steps 2 carried out incompletely), description of the reasons
Diagnosis of undernutrition and/or neurocognitive disorders and/or patent lung infection and/or COPD described in the patient's medical file, nutritional risk situation assessed by the Mini Nutritional Assessment® (MNA) | 19 months
  Patient characteristics will be collected at each site at the end of the study by a clinical research assistant based on their medical records.
Composition and disciplines of the care team | 19 months
  At the end of the study, all data on the each allied health professionals will be collected on the dysphaging sheet
Caregiver satisfaction (Likert scale). | 19 months
  At the end of the study, each allied health professionals who has been involved in the care of at least one patient will fill out a satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud - Court Séjour Gériatrique, Lyon, France

REFERENCES:
- [Derived] Durlach O, Tripoz-Dit-Masson S, Masse-Deragon N, Subtil F, Niasse-Sy Z, Herledan C, Guittard L, Goldet K, Merazga S, Chabert M, Suel A, Dayde D, Merdinian M, Falandry C. Feasibility of a screening and prevention procedure for risks associated with dysphagia in older patients in geriatric units: the DYSPHAGING pilot study protocol. BMJ Open. 2024 Apr 19;14(4):e081333. doi: 10.1136/bmjopen-2023-081333. PMID 38642998